CLINICAL TRIAL: NCT04112030
Title: Role of Digital Image Analysis in Diagnosing Nature of Indeterminate Biliary Duct Stricture
Brief Title: Role of DIA in Diagnosing Nature of Indeterminate Biliary Duct Stricture
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Abu Elfatth, Al-rahji University Hospital, Faculty of Medicine, Assiut, Egypt, Assiut University
Other Study IDs: DIA and biliary stricture
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Bile Duct Stricture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biliary brush sample were subjected to routine cytology and digital image analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Digital image analysis

SUMMARY:
The study aimed to assess role of DIA in diagnosing nature of indeterminate bile ducts stricture

DETAILED DESCRIPTION:
Biliary strictures (BSs) are common in clinical practice, but differentiating nature of the stricture either benign or malignant remains a challenge. Although there is a great advance in imaging and laboratory investigations, nature of BS is still unclear in some patients. Therefore, preoperative evaluation of such strictures is mandatory to put suitable plan with appropriate management.

BS is considered indeterminate biliary duct stricture (IBDS) if it has the following conditions; 1) no obvious mass on abdominal ultrasound (US), or magnetic resonance cholangiopancreatography (MRCP); 2) no distant metastasis on abdominal US, or MRI; and 3) no recent history of hepatobiliary surgery in the last 3 months.

IBDS has a particularly complex challenge, because patients and their physicians must weigh the malignant potential against benign etiologies in the face of morbidity of surgical intervention. About 15-24% of the patients had surgical intervention for suspected IBDS have a benign aetiology. Therefore, preoperative evaluation of such strictures is mandatory to put suitable plan with appropriate management.

Conventional cytological evaluation (CCE) has become the standard modality of practice for the investigation of such stricture. CCE had low diagnostic yield with an overall sensitivity of 41.6% and a negative predictive value of 58%. This low diagnostic yield is mainly attributed to desmoplastic reaction in BS.

Radiological elevation of BS with different modalities as MRCP enables us to detect the stricture and its extent and exclude other causes of obstruction. These modalities fail to determine nature of BS in many cases. In addition to, inability to take tissue sampling or perform therapeutic intervention.

Recently, there is a great advance in endoscopic assessment of BS as cholangioscopy, intraductal ultrasonography (IDUS), and confocal laser endomicroscopy. These techniques have high diagnostic yield in diagnosing nature of BS but secondary to high cost, complexity, and unavailability of these procedures, making them of limited use in evaluation the nature of IBDS.

Advanced cytological techniques have been emerged to identify nature of IBDS i.e., digital image analysis (DIA), and fluorescence in-situ hybridization (FISH) where both techniques detect the chromosomal alterations in malignant cells.

FISH is significantly more sensitive than CCE for assessment the nature of IBDS. However, the specificity of FISH was poor compared to the excellent specificity of CCE. The compromised specificity of FISH may limit its utility in the detection of nature of IBDS.

DIA has been widely used in many malignant diseases, especially in cervical cancer where it had 70% to 91.7%, sensitivity and 54.1% to 100% specificity for the diagnosis of different malignant diseases in published studies.

Role of DIA in pancreatobiliary malignancies is still controversial. Also, there are limited studies that have addressed the use of DIA in diagnosing the nature of IBDS. In addition to unavailability, the high cost and the complexity of advanced endoscopes, we designed this work to evaluate the diagnostic performance of DIA in identification nature of IBDS in comparison to CCE. Also, we perform a cost analysis of DIA vs. CCE in diagnosing nature of IBDS.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presented with biliary stricture with no obvious cause in abdominal imaging

Exclusion Criteria:

* biliary obstruction due to other causes as stones, or tumor,
* biliary surgery within the last six months
* Coagulopathy
* lost follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study included 50 patients with biliary stricture with no obvious cause in MRCP
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of DIA compared to routine cytology in case of IBDS | Baseline
  all samples were subjected to DIA and routine cytology and the result was compared with final diagnosis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JY, Jeon TJ. Factors Associated with Malignant Biliary Strictures in Patients with Atypical or Suspicious Cells on Brush Cytology. Clin Endosc. 2019 Mar;52(2):168-174. doi: 10.5946/ce.2018.105. Epub 2019 Jan 9. PMID 30625267
- [Background] Aljahdli ES. Management of distal malignant biliary obstruction. Saudi J Gastroenterol. 2018 Mar-Apr;24(2):71-72. doi: 10.4103/sjg.SJG_611_17. No abstract available. PMID 29637911
- [Derived] Helmy A, Saad Eldien HM, Seifeldein GS, Abu-Elfatth AM, Mohammed AA. Digital Image Analysis has an Additive Beneficial Role to Conventional Cytology in Diagnosing the Nature of Biliary Ducts Stricture. J Clin Exp Hepatol. 2021 Mar-Apr;11(2):209-218. doi: 10.1016/j.jceh.2020.07.009. Epub 2020 Jul 26. PMID 33746446